CLINICAL TRIAL: NCT07383324
Title: Impact of Indoor Overheating on Physiological Strain in Individuals With Schizophrenia
Brief Title: Heat Stress in Individuals With Schizophrenia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ottawa (Other)
Responsible Party: Principal Investigator, Glen P. Kenny, Full Professor, University Research Chair, University of Ottawa
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: HEPRU-2026-01-A
Record Dates: First submitted 2026-01-20; First posted 2026-02-03 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Heat Stress; Physiological Stress; Cognitive Change
Keywords: Indoor overheating; Indoor temperatures; Heat wave; Thermoregulation; Schizophrenia; Heat strain; Heat vulnerability; Hyperthermia; Mental health; Thermal comfort; Physical activity
MeSH Terms: conditions — Heat Stress Disorders; Schizophrenia; Hyperthermia; Psychological Well-Being; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exposure to indoor temperature upper limit of 26°C (Experimental): Participants exposed daylong (6 hours) to an indoor temperature maintained at 26°C and 45% relative humidity (humidex equivalent of 29).
  Interventions: Other: Simulated exposure to indoor overheating
- Exposure to hot indoor environment of 36°C (Experimental): Participants exposed daylong (6 hours) to an indoor temperature maintained at 36°C and 45% relative humidity (humidex equivalent of 45).
  Interventions: Other: Simulated exposure to indoor overheating

INTERVENTIONS:
Other: Simulated exposure to indoor overheating — Individuals with schizophrenia exposed to a 6-hour simulated heat exposure

SUMMARY:
Schizophrenia is a severe mental illness affecting approximately 24 million people worldwide and is associated with more than double the all cause mortality risk of the general population. Emerging evidence demonstrates that elevated temperatures acutely worsen mental health symptoms and significantly increase the risk of heat related morbidity and mortality. For people living with schizophrenia, prolonged exposure to heat can exacerbate psychiatric symptoms, impair judgment and decision making, and reduce the ability to engage in protective behaviors such as increasing hydration, reducing clothing, improving ventilation, or seeking cooler environments. As a result, individuals with schizophrenia may experience higher rates of heat related illness. To date our understanding of heat exposure effects in individuals with schizophrenia remains incomplete, hindering the development of evidence-based strategies to protect them.

Thus, the primary objective of this exploratory study is to gather preliminary data on the effects of indoor overheating on physiological responses (core body temperature and cardiovascular function), cognitive performance (attention, working memory, and reaction time), and mood in adults with schizophrenia. Specifically, we will assess whether maintaining indoor conditions at the upper recommended temperature limit for older adults (26°C, 45% relative humidity [RH]; PMID: 38329752) is sufficient to mitigate physiological strain compared with exposure to a hot indoor environment (36°C, 45% RH) representative of non-air-conditioned homes during extreme heat events in individuals with schizophrenia. In both conditions, the individual will remain seated at rest while wearing light clothing (t shirt and shorts), with the exception of performing 15 minutes of stepping exercise (4-4.5 METS) each hour (excluding the lunch period) to reflect typical daily activities of daily living.

ELIGIBILITY:
Inclusion Criteria:

* English or French speaking.
* Ability to provide informed consent.
* Individuals with and without schizophrenia or schizoaffective disorder.

Exclusion Criteria:

* Endurance exercise training (greater than 3 sessions of vigorous exercise training per week for 30 minutes or more)
* Restrictions to physical activity
* Any history of diagnoses for other psychiatric disorders deemed to make participation in the study inadvisable.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-11-08 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Core temperature (Peak) during daylong exposure to indoor overheating | End of 6 hour daylong exposure
  Peak visceral temperature (15 min average) during exposure. Visceral temperature is measured continuously throughout the 6 hour exposure to the simulated indoor overheating.
Core temperature (AUC) during daylong exposure to indoor overheating | End of 6 hour daylong exposure
  Areas under the curve (AUC) of visceral temperature during the 6 hour exposure to the simulate indoor overheating.
Core temperature end of daylong exposure to indoor overheating | End of 6 hour daylong exposure
  Visceral temperature measured at hour 6 of exposure to indoor overheating (15-min average).
Mean skin temperature (Peak) during daylong exposure to indoor overheating | End of 6 hour daylong exposure
  Peak mean skin temperature (15 min average) during exposure. Mean skin temperature as calculated from skin temperature measured across 7 body regions is measured continuously throughout the 6 hour exposure to the simulated indoor overheating.
Mean skin temperature (AUC) during daylong exposure to indoor overheating | End of 6 hour daylong exposure
  Areas under the curve (AUC) of mean skin temperature as calculated over 7 body regions during the 6 hour exposure to the simulate indoor overheating.
Mean skin temperature end of daylong exposure to indoor overheating | End of 6 hour daylong exposure
  Mean skin temperature measured over 7 body regions at hour 6 of exposure to indoor overheating (15-min average).
Heat rate (Peak) during daylong exposure to indoor overheating | End of 6 hour daylong exposure
  Peak heart rate (15 min average) during exposure. Heart rate is measured continuously throughout the 6 hour exposure to the simulated indoor overheating.
Heart rate (AUC) during daylong exposure to indoor overheating | End of 6 hour daylong exposure
  Areas under the curve (AUC) of heart rate during the 6 hour exposure to the simulate indoor overheating.
Heart rate end of daylong exposure to indoor overheating | End of 6 hour daylong exposure
  Heart rate measured at hour 6 of exposure to indoor overheating (15-min average).
Systolic blood pressure during daylong exposure to indoor overheating | At the start (hour 0) and end of 6 hour daylong exposure
  Systolic blood pressure measured in triplicate via automated oscillometry (~60 seconds between measures).
Diastolic blood pressure during daylong exposure to indoor overheating. | At the start (hour 0) and end of 6 hour daylong exposure
  Diastolic blood pressure measured in triplicate via automated oscillometry (~60 seconds between measures).
Reaction time during daylong exposure to indoor overheating (cognitive function). | At the start (hour 0) and end of 6 hour daylong exposure
  Participants will be provided with a tablet device with the Sway Medical testing platform for the assessment of reaction time. Participants will be asked to initiate a movement of the device in response to a visual cue.
Impulse control during daylong exposure to indoor overheating (cognitive function). | At the start (hour 0) and end of 6 hour daylong exposure
  Participants will be provided with a tablet device with the Sway Medical testing platform for the assessment of impulse control. Participants will be asked to respond to both "go" and "no-go" visual cues. In response to the "go" cue, participants will initiate a movement of the device.
Memory recall during daylong exposure to indoor overheating (cognitive function). | At the start (hour 0) and end of 6 hour daylong exposure
  Participants will be provided with a tablet device with the Sway Medical testing platform for the assessment of memory recall. Participants complete both a delayed recall test and a working memory test.
CDC 4-Stage Balance Test during daylong exposure to indoor overheating (postural stability). | At the start (hour 0) and end of 6 hour daylong exposure
  To assess postural stability, participants hold a tablet to their chest, then auditory cues guide participants through four consecutive stances, feet side by side, instep of one foot touching the big toe of the other foot, tandem stand with one foot in front of the other, heel touching toe, and stand on one foot. The balance assessment will be evaluated based on movement detected by an accelerometer integrated into the hardware of the tablet device (Sway Medical Inc).
Executive function during daylong exposure to indoor overheating (cognitive function). | At the start (hour 0) and end of 6 hour daylong exposure
  Participants will be provided with a tablet device with the Sway Medical testing platform for the assessment of executive function. Participants will complete the Cued Stroop test, in which they are presented a sequence of congruent, neutral and incongruent color-word tasks.
BTrackS Balance Assessment during daylong exposure to indoor overheating (postural stability). | At the start (hour 0) and end of 6 hour daylong exposure
  To assess postural stability, participants will be asked to stand on a BTracks force plate with their feet spread out to shoulder width, hand on their hips and eyes closed. The assessment will comprise of four trials (one practice trial) lasting 20 seconds in length and 20 seconds between trials. Center of pressure (COP) vector data along vertical (y) and horizontal (x) axes will be summed for the total path excursion length (cm) during each trial
Hydration status during daylong exposure to indoor overheating | At the start (hour 0) and end of 6 hour daylong exposure
  Hydration status measured via assessing the urine specific gravity of a urine sample.
Fluid consumption during daylong exposure to indoor overheating | At end of 6 hour daylong exposure
  Average hourly fluid consumption calculated by weighing participant water intake at the start and end of each hour of exposure (normalized to the exposure duration).
Fluid loss during daylong exposure to indoor overheating | At end of 6 hour daylong exposure
  Fluid loss calculated as the change in body mass during each exposure presented as a percentage of baseline body mass (corrected for food consumption).
Thermal sensation scale during daylong exposure to indoor overheating | At the start (hour 0) and end of 6 hour daylong exposure
  Thermal sensation assessed via an ordinal scale (How hot do you feel?) ranging from "extremely hot" to "neutral".
Thermal sensation 2 scale during daylong exposure to indoor overheating | At the start (hour 0) and end of 6 hour daylong exposure
  Thermal sensation assessed via an ordinal scale ("How do you feel?") ranging from "hot" to "cold" (midpoint: neutral)
Thermal comfort scale during daylong exposure to indoor overheating | At the start (hour 0) and end of 6 hour daylong exposure
  Thermal comfort assessed via an ordinal scale ("How comfortable does your body temperature feel?") ranging from "very uncomfortable" to "comfortable".
Thirst sensation scale during daylong exposure to indoor overheating | At the start (hour 0) and end of 6 hour daylong exposure
  Thirst sensation assessed via an ordinal scale ranging from very, very thirsty to not thirsty at all.
Feel good scale during daylong exposure to indoor overheating | At the start (hour 0) and end of 6 hour daylong exposure
  Feel good scale assessed via an ordinal scale (How good do you feel?) ranging from "very good" to "very bad" (midpoint: neutral)
Activity levels (total steps taken) during daylong exposure to indoor overheating | End of 6 hour daylong exposure
  Activity levels, quantified by number of steps taken per hour and totaled for each 6 hour exposure, assessed via a wearable accelerometer worn on the wrist and hip.
Perceived exertion scale during daylong exposure to indoor temperature limit. | At the start (hour 0) and end of 6 hour daylong exposure
  Perceived exertional assessed via an ordinal scale ("How hard are you working?") ranging from "no exertional at all" to "maximal exertion"

SECONDARY OUTCOMES:
Profiles of Mood States (POMS) during daylong exposure to indoor overheating | At the start (hour 0) and end of 6 hour daylong exposure
  Potential changes in mood (7 subscales of mood: tension, anger, depression, fatigue, confusion, vigor and esteem related affect). The POMS-40 is a validated, self-administered questionnaire that examines seven distinct aspects of mood state across two positive subscales (Esteem-Related Affect, and Vigor) and five negative subscales (Fatigue, Tension, Confusion, Anger, and Depression), which are described across 40 distinct adjectives. For each individual item, participants are asked to describe "how you feel right now" by responding using a 5-point Likert scale (0 = "Not at all", 1 = "A little", 2 = "Moderately", 3 = "Quite a lot", or 4 = "Extremely"). The values of items associated with a specific subscale (e.g., Fatigue) are summed to calculate its score.
Environmental Symptoms Questionnaire (ESQ) during daylong exposure to indoor overheating | At the start (hour 0) and end of 6 hour daylong exposure
  Self-reported environmental reactions and medical symptomatology associated with prolonged heat exposure. The ESQ-IV is a validated 68-item, self-administered questionnaire that has been used successfully in identifying symptomatology during exposure to a wide variety of environmental conditions, including heat exposure. Participants are asked to assess and described "how you have been feeling today" by responding to each item using a 6-point Likert scale (0 = "Not at all", 1 = "Slight", 2 = "Somewhat", 3 = "Moderate", 4 = "Quite a bit", or 5 = "Extreme"). Total Symptom Score is calculated from this data by taking the sum of the intensity ratings from all 68 individual items using reverse scores for the three positive items from the list ("I Felt Good", "I Felt Alert", and "I Felt Wide Awake").

CONTACTS AND LOCATIONS:
Overall Officials: Glen P Kenny, PhD, Principal Investigator — University of Ottawa
Locations (1):
- University of Ottawa, Ottawa, Ontario, Canada